CLINICAL TRIAL: NCT02912455
Title: Canagliflozin vs. Placebo for Post Bariatric Patients With Persistent Type 2 Diabetes
Brief Title: CARAT: Canagliflozin vs. Placebo for Post Bariatric Patients With Persistent Type 2 Diabetes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was terminated due to difficulty with reaching enrollment goals
Sponsor: The Cleveland Clinic (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Sangeeta Kashyap, Associate Professor of Medicine, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-574
Record Dates: First submitted 2016-08-24; First posted 2016-09-23 (Estimated); Results first posted 2020-06-30 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
Keywords: Post-Bariatric Surgery; hemoglobin A1c protein, human
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Drug (canagliflozin) (Active Comparator): Subjects randomized to study drug will be assigned a six month course starting on canagliflozin 100 mg for two weeks titrated up to 300 mg daily (n= 24).
  Interventions: Drug: canagliflozin
- Placebo (Placebo Comparator): Subjects randomized to placebo will be assigned a six month course of one placebo pill daily (n =12).
  Interventions: Drug: Placebo (for canagliflozin)

INTERVENTIONS:
Drug: canagliflozin — encapsulated (gelatin capsule).
  Other Names: Invokana
  Arms: Study Drug (canagliflozin)
Drug: Placebo (for canagliflozin) — encapsulated (gelatin capsule). The placebo capsule filler is called micro-crystalline cellulose.
  Arms: Placebo

SUMMARY:
This is a prospective, randomized clinical trial for patients with recurrent type 2 diabetes post-gastric bypass surgery that will compare a 6 month course of canagliflozin monotherapy vs. placebo on clinical outcomes of type 2 diabetes.

DETAILED DESCRIPTION:
Following consent and a screening visit to assess eligibility and clinical status (i.e. historical, physical and biochemical parameters including glycemic control and a pregnancy test in females), a baseline visit with diabetes educator will take place to provide standard diabetes education, nutrition and exercise prescription.

Nutritional assessment for vitamin/mineral deficiency will be performed per clinical care guidelines at the screening visit. Subjects will be asked to take nutritional supplements (i.e. vitamins and minerals) per current clinical guidelines for post-bariatric patients. Stable doses of supplements will be established for at least 2 weeks prior to randomization. Thirty-six subjects with recurrent diabetes that are naïve to hypoglycemic agents with HbA1c greater than or equal to 6.5% and less than 10% will be randomly assigned to a six month course of a) canagliflozin 100mg for 2 weeks titrated up to 300 mg daily (N = 24) vs. placebo (n= 12) at the randomization. Patients taking an anti-diabetic medication will be asked to wash out for 8 weeks prior to the randomization visit. At randomization, biochemical assessment of glycemic parameters (fasting glucose, HbA1c), lipid panel, complete metabolic panel, uric acid, leptin, total and HMW adiponectin, C-reactive protein and urine for albumin/creatinine ratio will be performed. Dual-energy x-ray absorptiometry (DXA) scan will be performed for body fat composition.

Following randomization, subjects will be clinically evaluated at three office visits at 6 weeks, 3 and 6 months by PI and/or the research staff. The primary outcome measures at 6 months post-randomization include HbA1c followed by the change in HbA1c from randomization. Secondary measures include fasting glucose, BMI, change in body weight, blood pressure, lipid profile. Symptomatic hypoglycemia (blood glucose < 70) and drug related side effects (i.e. mycotic genital infections, urinary tract infection) will be monitored with adverse event reporting. Metabolic testing in all subjects at randomization and at 6 months will include a DXA scan for body fat composition and blood for leptin and adiponectin levels.

Rescue glucose lowering therapy will be provided for the control group for blood glucose >250 mg/dl. If chronic uncontrolled hyperglycemia (HbA1c >10%) occurs then basal bolus insulin will be implemented.

ELIGIBILITY:
Inclusion Criteria:

* Post Roux-n-Y gastric bypass (RYGB) surgery and sleeve gastrectomy (SG) patients who underwent surgery >1 and <15 years ago in the Cleveland surrounding area
* Age 20-75 years of age
* Type II Diabetes Mellitus (D2M) diagnosis (history, medication usage, biochemical criteria) prior to and after surgery; after surgery, defined by a single HbA1c of greater or equal to 6.5% at consent and screening.
* Metformin patients must have an HbA1c greater than or equal to 6.5% but less than or equal to 10% at randomization; for diet controlled patients (i.e. not on any T2D medication), HbA1c must be greater than or equal to 6.5% at randomization.
* Patient reporting of improvement in T2D status or objective improvements in T2D status at any time post-surgery.
* estimated glomerular filtration rate (eGFR) ≥ 60mL/min prior to randomization
* Has the ability and willingness to provide informed consent.
* Is able to understand the options and to comply with the requirements of each program
* Female subject agrees to have a serum pregnancy test at screening. A negative serum pregnancy test result is required prior to randomization.
* Female patients must agree to use a reliable method of contraception for 6 months or duration of intervention
* Patients taking an anti-diabetic medication, except insulin, are eligible and must agree to washout for 8 weeks prior to the randomization visit.

Exclusion Criteria:

* Type 1 diabetes indicated by history of diabetic ketoacidosis and lack of remission in response to bariatric surgery
* Other post bariatric procedures (banding, duodenal switch, biliopancreatic diversion)
* Current use of insulin.
* End organ diabetic complications (renal failure, cardiomyopathy, severe neuropathy/foot ulcers)
* Documented severe or unstable depression/anxiety or eating disorder that would not enable patient to adhere to anti-diabetic treatment
* Clinical contraindications to use canagliflozin, i.e., history of bladder cancer, Child-Pugh class C

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta Kashyap, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Drug (Canagliflozin): Subjects randomized to study drug will be assigned a six month course starting on canagliflozin 100 mg for two weeks titrated up to 300 mg daily (n= 11).
  canagliflozin: encapsulated (gelatin capsule).
- Placebo: Subjects randomized to placebo will be assigned a six month course of one placebo pill daily (n =5).
  Placebo (for canagliflozin): encapsulated (gelatin capsule). The placebo capsule filler is called micro-crystalline cellulose.
Period: Overall Study
Arm/Group | Study Drug (Canagliflozin) | Placebo
Started | 11 | 5
Completed | 9 | 2
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Study Drug (Canagliflozin): Subjects randomized to study drug will be assigned a six month course starting on canagliflozin 100 mg for two weeks titrated up to 300 mg daily.
  canagliflozin: encapsulated (gelatin capsule).
- Placebo: Drug: Placebo (for canagliflozin)
  encapsulated (gelatin capsule). The placebo capsule filler is called micro-crystalline cellulose.
- Total: Total of all reporting groups
Arm/Group | Study Drug (Canagliflozin) | Placebo | Total
Number analyzed (Participants) | 11 | 5 | 16
Age, Continuous [Median (Full Range); unit: years] | 58 [38 to 75] | 44.0 [34.0 to 59.0] | 54.0 [34.0 to 75.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 4 | 1 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11 | 5 | 16
BMI [Median (Full Range); unit: kg/m^2] | 39.6 [28.6 to 49.4] | 37.9 [31.9 to 44.7] | 39.2 [28.6 to 49.4]
Height (m) [Median (Full Range); unit: meters] | 1.7 [1.5 to 1.7] | 1.7 [1.6 to 1.9] | 1.7 [1.5 to 1.9]
Weight (kg) [Median (Full Range); unit: kg] | 108.6 [78.3 to 132.9] | 117.5 [86.0 to 133.7] | 108.9 [78.3 to 133.7]
Hemoglobin A1c (%) [Median (Full Range); unit: percent] | 7.2 [6.5 to 8.3] | 8.2 [6.9 to 10.0] | 7.4 [6.5 to 10.0]
Fasting glucose (mg/dL) [Median (Full Range); unit: mg/dL] | 163.0 [105.0 to 204.0] | 164.0 [116.0 to 239.0] | 163.5 [105.0 to 239.0]
Diastolic blood pressure (mm/Hg) [Median (Full Range); unit: mmHg] | 73.0 [52.0 to 87.0] | 77.0 [51.0 to 86.0] | 76.5 [51.0 to 87.0]
Systolic blood pressure (mm/Hg) [Median (Full Range); unit: mmHg] | 137.0 [106.0 to 148.0] | 133.0 [117.0 to 141.0] | 134.5 [106.0 to 148.0]
Uric acid (mg/dL) [Median (Full Range); unit: mg/dL] | 4.9 [2.9 to 7.9] | 3.9 [3.3 to 5.1] | 4.3 [2.9 to 7.9]
Total cholesterol (mg/dL) [Median (Full Range); unit: mg/dL] | 160.0 [112.0 to 257.0] | 167.0 [135.0 to 202.0] | 162.0 [112.0 to 257.0]
Triglycerides (mg/dL) [Median (Full Range); unit: mg/dL] | 130.0 [59.0 to 224.0] | 107.0 [62.0 to 121.0] | 109.5 [59.0 to 224.0]
LDL (mg/dL) [Median (Full Range); unit: mg/dL] | 87.0 [31.0 to 175.0] | 108.0 [67.0 to 120.0] | 92.0 [31.0 to 175.0]
HDL (mg/dL) [Median (Full Range); unit: mg/dL] | 47.0 [28.0 to 81.0] | 51.0 [29.0 to 60.0] | 49.0 [28.0 to 81.0]
Body fat % [Median (Full Range); unit: percentage of body fat] | 49.3 [30.5 to 55.3] | 44.1 [29.4 to 51.0] | 48.6 [29.4 to 55.3]
Lean mass % [Median (Full Range); unit: percentage of lean mass] | 50.7 [44.7 to 69.5] | 55.9 [49.0 to 70.6] | 51.5 [44.7 to 70.6]
Truncal fat [Median (Full Range); unit: percentage of truncal fat] | 53.5 [36.8 to 55.3] | 47.8 [34.9 to 54.0] | 50.9 [34.9 to 55.3]
Android fat [Median (Full Range); unit: percentage of android fat] | 55.6 [41.1 to 58.6] | 51.3 [38.0 to 56.3] | 53.9 [38.0 to 58.6]
Gynoid fat [Median (Full Range); unit: percentage of gynoid fat] | 48.1 [27.5 to 55.3] | 47.3 [30.1 to 55.6] | 47.7 [27.5 to 55.6]
Spine BMD [Median (Full Range); unit: g/cm^2] | 1.2 [1.03 to 1.8] | 1.3 [1.05 to 1.3] | 1.2 [1.03 to 1.8]
Leg BMD [Median (Full Range); unit: g/cm^2] | 1.2 [1.07 to 1.9] | 1.2 [1.05 to 1.4] | 1.2 [1.05 to 1.9]
HMW adiponectin [Median (Full Range); unit: ug/mL] | 2.9 [0.8 to 10] | 3.3 [1.6 to 7] | 3.1 [0.8 to 10]
Adiponectin [Median (Full Range); unit: ug/mL] | 4.2 [1.5 to 17] | 5 [3 to 10] | 4.6 [1.5 to 17]
Leptin [Median (Full Range); unit: ng/mL] | 28 [5.3 to 87] | 29 [4.7 to 117] | 28.5 [4.7 to 117]
CRP [Median (Full Range); unit: mg/L] | 4.1 [1.00 to 44.5] | 0.45 [0.20 to 3.8] | 3.7 [0.20 to 44.5]

OUTCOME MEASURES:

1. Primary Outcome: Change at Six Months Versus Baseline in Hemoglobin A1c Value (%)
Description: The change in hemoglobin A1c from randomization following the 6 month administration of canagliflozin vs. placebo in patients with type 2 diabetes post-bariatric surgery
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Study Drug (Canagliflozin) | Placebo
Number analyzed (Participants) | 11 | 5
percentage | -0.31 [-0.72 to 0.10] | 0.11 [-0.71 to 0.93]

2. Secondary Outcome: Change in Fasting Glucose From Randomization
Description: The change in fasting glucose from randomization following the 6 month administration of canagliflozin vs. placebo in patients with type 2 diabetes post-bariatric surgery.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Study Drug (Canagliflozin) | Placebo
Number analyzed (Participants) | 11 | 5
mg/dL | -32.90 [-56.02 to -9.79] | -44.61 [-102.39 to 13.17]

3. Secondary Outcome: Change in Body Weight at Six Months Compared to Baseline
Description: The change in body weight from randomization following the 6 month administration of canagliflozin vs. placebo in patients with type 2 diabetes post-bariatric surgery.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Study Drug (Canagliflozin) | Placebo
Number analyzed (Participants) | 11 | 5
kilograms | -3.77 [-6.33 to -1.22] | 6.33 [-1.50 to 14.16]

4. Secondary Outcome: Change in Total Cholesterol
Description: The change in total cholesterol from randomization following the 6 month administration of canagliflozin vs. placebo in patients with type 2 diabetes post-bariatric surgery
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Study Drug (Canagliflozin) | Placebo
Number analyzed (Participants) | 11 | 5
mg/dL | -0.87 [-26.59 to 24.85] | 3.69 [-37.53 to 44.92]

5. Secondary Outcome: Change in Diastolic Blood Pressure at Six Months Compared to Baseline
Description: The change in diastolic blood pressure from randomization following the 6 month administration of canagliflozin vs. placebo in patients with type 2 diabetes post-bariatric surgery
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Study Drug (Canagliflozin) | Placebo
Number analyzed (Participants) | 11 | 5
mmHg | -1.18 [-6.62 to 4.26] | 2.95 [-13.69 to 19.60]

6. Secondary Outcome: Change in Adiponectin Levels at 6 Months Compared to Randomization
Description: The change in adiponectin levels from randomization following the 6 month administration of canagliflozin vs. placebo in patients with type 2 diabetes post-bariatric surgery.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Study Drug (Canagliflozin) | Placebo
Number analyzed (Participants) | 11 | 5
ug/mL | 0.7 [-2.2 to 5.7] | -3.4 [-9.3 to 2.5]

7. Secondary Outcome: Change in Leptin Levels at 6 Months Compared to Baseline
Description: Change in leptin levels at 6 months compared to baseline The change in leptin levels from randomization following the 6 month administration of canagliflozin vs. placebo in patients with type 2 diabetes post-bariatric surgery.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Study Drug (Canagliflozin) | Placebo
Number analyzed (Participants) | 11 | 5
ng/mL | -8.1 [-35.1 to 18.9] | -11 [-93.1 to 71.1]

8. Secondary Outcome: Change in CRP Levels at 6 Months Compared to Baseline
Description: The change in C-reactive protein levels from randomization following the 6 month administration of canagliflozin vs. placebo in patients with type 2 diabetes post-bariatric surgery.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Study Drug (Canagliflozin) | Placebo
Number analyzed (Participants) | 11 | 5
mg/L | -5.35 [-13.81 to 3.12] | 3.34 [-0.76 to 7.44]

9. Secondary Outcome: Number of Participants Who Reported Hypoglycemia From Each Group (at a Frequency of 1 Episode)
Description: The number of participants who reported symptomatic hypoglycemia episodes from randomization following the 6 month administration of canagliflozin vs. placebo in patients with type 2 diabetes post-bariatric surgery.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Study Drug (Canagliflozin) | Placebo
Number analyzed (Participants) | 11 | 5
participants | 2 | 0

10. Secondary Outcome: Change in Percent Body Fat as Measured by DEXA Scan at 6 Months Compared to Randomization
Description: The change in body fat from randomization following the 6 month administration of canagliflozin vs. placebo in patients with type 2 diabetes post-bariatric surgery.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Study Drug (Canagliflozin) | Placebo
Number analyzed (Participants) | 11 | 5
percent change | -1.82 [-3.83 to 0.20] | 2.65 [-1.21 to 6.51]

11. Secondary Outcome: Change in Systolic Blood Pressure at 6 Months Compared to Baseline
Description: The Change in Systolic Blood Pressure From Randomization Following the 6 Month Administration of Canagliflozin vs. Placebo in Patients With Type 2 Diabetes Post-bariatric Surgery
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Study Drug (Canagliflozin) | Placebo
Number analyzed (Participants) | 11 | 5
mmHg | 4.62 [-7.10 to 16.34] | 12.63 [-5.02 to 30.28]

12. Secondary Outcome: Change in Percentage of Lean Mass
Description: Change in percentage of lean body mass as measured by DEXA scan at 6 months compared to randomization
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Study Drug (Canagliflozin) | Placebo
Number analyzed (Participants) | 11 | 5
percent change | 1.82 [-0.20 to 3.83] | -2.65 [-6.51 to 1.21]

13. Secondary Outcome: Change in Percentage of Truncal Fat
Description: Change in percentage of truncal fat as measured by DEXA scan at 6 months compared to randomization
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Study Drug (Canagliflozin) | Placebo
Number analyzed (Participants) | 11 | 5
percent change | -2.67 [-5.19 to -0.16] | 2.74 [-0.14 to 5.63]

14. Secondary Outcome: Change in Percentage of Android Fat
Description: Change in percentage of android fat as measured by DEXA scan at 6 months compared to randomization
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Study Drug (Canagliflozin) | Placebo
Number analyzed (Participants) | 11 | 5
percent change | -3.00 [-5.67 to -0.32] | 3.33 [0.23 to 6.43]

15. Secondary Outcome: Change in Percentage of Gynoid Fat
Description: Change in percentage of gynoid fat as measured by DEXA scan at 6 months compared to randomization
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Study Drug (Canagliflozin) | Placebo
Number analyzed (Participants) | 11 | 5
percent change | -1.69 [-3.65 to 0.28] | 2.17 [-2.26 to 6.59]

16. Secondary Outcome: Change in Spine Bone Mineral Density
Description: Change in spine bone marrow density as measured by DEXA scan at 6 months compared to randomization
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: grams per square centimeter
Arm/Group | Study Drug (Canagliflozin) | Placebo
Number analyzed (Participants) | 11 | 5
grams per square centimeter | -0.02 [-0.07 to 0.03] | 0.14 [-0.11 to 0.40]

17. Secondary Outcome: Change in Leg Bone Mineral Density
Description: Change in leg bone marrow density as measured by DEXA scan at 6 months compared to randomization
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: grams per square centimeter
Arm/Group | Study Drug (Canagliflozin) | Placebo
Number analyzed (Participants) | 11 | 5
grams per square centimeter | 0.01 [-0.03 to 0.05] | -0.04 [-0.37 to 0.28]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 6 months.
Arm/Group | Study Drug (Canagliflozin) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/5
Other Adverse Events (participants affected / at risk) | 7/11 | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Drug (Canagliflozin) (N=11) | Placebo (N=5)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (8) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Increased thirst (Metabolism and nutrition disorders) | 5 (6) | 2 (2)
Increased urination (Metabolism and nutrition disorders) | 5 (6) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1)
Genital yeast infection (Renal and urinary disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lightheadedness (Nervous system disorders) | 2 (2) | 0 (0) — Vertigo/Dizziness
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased hunger (Investigations) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT02912455/Prot_SAP_000.pdf